CLINICAL TRIAL: NCT02449434
Title: Timing of Dietary Acid Intake, Brushing Teeth and Acid Erosion.
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: RJ114/N205
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2016-02

CONDITIONS: Tooth Wear
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Severe Tooth Wear: Severe tooth wear with a BEWE score of 12 and at least one score of 3 in three quadrants Adult 18 years or older No missing anterior teeth Minimum of at 10 teeth in the upper and 10 teeth in the lower jaw No anterior crowns/ bridges or implants Written consent to the study
  There was no intervention - just a questionnaire for each group
- Without Tooth Wear: BEWE score of 10 or lower and no score of 3 on any surface of any tooth (clinically classified as no or mild erosive tooth wear) Adult 18 years or older No missing anterior teeth Minimum of at 10 teeth in the upper and 10 teeth in the lower jaw No anterior crowns/ bridges or implants Written consent to the study
  There was no intervention - just a questionnaire for each group

SUMMARY:
This is a questionnaire based study investigating the relationship between the timing of dietary acid intake toothbrushing and erosive tooth wear. Data will be collected on the timing, nature, frequency and duration of dietary acid intakes and timing and frequency of the participants toothbrushing. Signs of the participants erosive tooth wear will then be recorded

DETAILED DESCRIPTION:
The study group will consist of two cohorts, those presenting with tooth wear and a control group. Participants will be recruited from the care planning clinic of the Dental Institute King's College London. Suitable participants meeting the inclusion criteria will be approached on the clinic, given the patient information sheet and asked to consider participating. Written consent will be obtained from those accepting the request. An interviewer-led, previously validated questionnaire will question their frequency and timing of dietary acid intake, tooth brushing and any habits associated with dietary acid intake. This will be followed by a Basic Erosive Wear Examination.

The process will take 7-8 minutes and the participant is free to withdraw at any time

ELIGIBILITY:
Inclusion Criteria:

1. Severe tooth wear with a BEWE score of 12 and at least one score of 3 in three quadrants
2. Adult 18 years or older
3. No missing anterior teeth
4. minimum of at 10 teeth in the upper and 10 teeth in the lower jaw
5. No anterior crowns/ bridges or implants
6. Written consent to the study

Exclusion Criteria:

1. Pregnancy
2. Participation in other research within 30 days
3. Unable to speak or understand English
4. Presence of periodontal disease or caries on more than one tooth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred into the Dental institute of King's College London for dental treatment
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bartlett, BDS PhD, Principal Investigator — King's College London
Locations (1):
- Dental Institute, Guy's Hospital, London, United Kingdom

REFERENCES:
- [Result] O'Toole S, Bernabe E, Moazzez R, Bartlett D. Timing of dietary acid intake and erosive tooth wear: A case-control study. J Dent. 2017 Jan;56:99-104. doi: 10.1016/j.jdent.2016.11.005. Epub 2016 Nov 14. PMID 27856311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (n = 600) aged 18 years or older, were recruited between May 2014 and March 2016 following referral by their general dental practitioners (GDP) for erosive tooth wear (cases, n = 300) or general treatment (controls, n = 300) to the restorative clinics at King's College London Dental Institute.
Groups:
- Severe Erosive Tooth Wear: a BEWE score of 12 or higher and at least one score of 3 in a sextant
- Mild/Moderate Erosive Tooth Wear: A BEWE score of 10 or lower and no score of 3 on any surface of any tooth
Period: Overall Study
Arm/Group | Severe Erosive Tooth Wear | Mild/Moderate Erosive Tooth Wear
Started | 300 | 300
Completed | 300 | 300
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Severe Erosive Tooth Wear: BEWE score of 12 or higher and at least one score of 3 in a sextant whereas
- Mild/Moderate Erosive Tooth Wear: BEWE score of 10 or lower and no score of 3 on any surface of any tooth
- Total: Total of all reporting groups
Arm/Group | Severe Erosive Tooth Wear | Mild/Moderate Erosive Tooth Wear | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 285 | 285 | 570
  >=65 years | 15 | 15 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 175 | 313
  Male | 162 | 125 | 287
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 300 | 300 | 600

OUTCOME MEASURES:

1. Primary Outcome: Basic Erosive Wear Examination
Description: Each tooth will be graded by the extent of the surface which the acid has damaged. The Basic Erosive Wear Examination (BEWE) index will grade tooth wear on the buccal, occlusal and palatal/lingual surfaces of each tooth excluding third molars. This ordinal scale graded tooth wear from 0 to 3 (0 = no wear, 1 = early surface loss, 2 = surface loss < 50% or specific defect, 3 = surface loss > 50%). The worst score in each sextant will be taken to be the sextant score. A cumulative score will be calculated for the mouth by adding each sextant score, which can range from 0-18. A higher score indicates a higher level of erosive tooth wear (worse outcome)
Time Frame: Single reading of wear of the teeth at the appointment date. Examination of wear takes 5 minutes
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Severe Erosive Tooth Wear: Erosive tooth wear cases were defined as those with a BEWE score of 12 or higher and at least one score of 3 in a sextant
- Mild/Moderate Erosive Tooth Wear: Controls were defined as those with a BEWE score of 10 or lower and no score of 3 on any surface of any tooth (clinically classified as no or mild erosive tooth wear)
Arm/Group | Severe Erosive Tooth Wear | Mild/Moderate Erosive Tooth Wear
Number analyzed (Participants) | 300 | 300
Units on a scale | 15.01 (2.3) | 6.27 (2.79)
Statistical Analysis 1: Comparison: Severe Erosive Tooth Wear vs Mild/Moderate Erosive Tooth Wear; A minimum sample size of 490 participants (245 in each group) was needed. This calculation assumed the proportion of adults with high dietary acid intake (3+ times/day) was 55% among cases and 40% among controls (expected odds ratio of 2.25), case- control ratio of 1-to-1, 90% statistical power and 95% significance level; Test type: Other — Using the presence or absence of severe erosive wear as the dependent variable, the unadjusted, sex-and-age- adjusted and fully adjusted associations of the included variables with erosive tooth wear were estimated using unconditional binary logistic regression and reported using odds ratios (OR); p < 0.05, Regression, Logistic — Only results from fully adjusted regression models will be deemed as significant; Unconditional binary logistic regression and reported using odds ratios and 95% confidence intervals; Odds Ratio (OR) = 2.25

ADVERSE EVENTS:
Time Frame: Non applicable -- All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: Non applicable -- All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Groups:
- Severe Erosive Tooth Wear: BEWE score of 12 or higher and at least one score of 3 in a sextant
  Non applicable -- All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
- Mild/Moderate Erosive Tooth Wear: BEWE score of 10 or lower and no score of 3 on any surface of any tooth
  Non applicable -- All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Severe Erosive Tooth Wear | Mild/Moderate Erosive Tooth Wear
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-12-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT02449434/Prot_SAP_000.pdf
  • Informed Consent Form (2013-12-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT02449434/ICF_001.pdf